CLINICAL TRIAL: NCT02784990
Title: Study of Pancreatic Enzymes in the Drains as Early Biomarkers of Post-operative Pancreatic Fistula and Its Clinical Repercussions
Acronym: LIPA-DRAIN
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: FACY PHRCI 2015
Record Dates: First submitted 2016-05-18; First posted 2016-05-27 (Estimated); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Pancreatic Fistula
MeSH Terms: conditions — Pancreatic Fistula | interventions — Lipase; Amylases; C-Reactive Protein

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patient
  Interventions: Biological: Lipase, amylase and CRP (C-reactive protein) dosages

INTERVENTIONS:
Biological: Lipase, amylase and CRP (C-reactive protein) dosages

SUMMARY:
Surgery is the principal treatment for benign and malignant pancreatic tumours. This surgery can be accompanied by complications among which the main one is pancreatic fistula, which leads to the flow of pancreatic juices into the abdominal cavity. Depending on its severity, a fistula can be managed medically, with the implantation of a la pose d'un percutaneous drain, endoscopic treatment, or revisit surgery. It has been shown that early management of the fistula prevents it from evolving towards major complications such as haemorrhage or serious intra-abdominal infections.

To date, the early diagnosis of pancreatic fistula is based on high levels of one pancreatic enzyme, amylase, in the drains. However in certain clinical situations, patients present post-operative fistulas with no elevation of amylase. And, on the contrary, increased amylase with no clinical consequences.

It is therefore necessary to identify another early early marker of pancreatic fistula that corresponds better to clinical signs.

In a preliminary study conducted in 65 patients, the investigators recently found that another pancreatic enzyme (lipase) could be a more pertinent marker of pancreatic fistula, but this requires confirmation in a greater number of patients.

The objective is to evaluate the diagnostic performance of lipase in the drains for the early detection of pancreatic fistula with clinical repercussions in the 30 days following the surgery.

The study consists in collecting at 4 different time points (D1, D3, D4 and D6) a tube of blood and a tube of drain liquid.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18
* Patients undergoing scheduled pancreatic resection with or without anastomosis (cephalic duodenopancreatectomy, median pancreatectomy, left pancreatectomy, enucleation)
* Patients able to understand instructions/information
* Patients who have provided written informed consent
* Patients with Health Insurance cover

Exclusion Criteria:

* Patients with scheduled total pancreatectomy
* Adults under wardship
* Pregnant or breast-feeding women
* Total pancreatectomy
* Pancreatectomy not feasible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing scheduled pancreatic resection
Sampling Method: Non-Probability Sample
Enrollment: 770 (Actual)
Dates: Start 2016-06-03 (Actual); Primary Completion 2020-11-03 (Actual); Study Completion 2020-11-03 (Actual)

PRIMARY OUTCOMES:
Dosage of lipase in the drains | 3 days after surgical resection

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - CHU Jean Minjoz, Besançon
  - CHU William MOREY, Chalon-sur-Saône
  - CHU Dijon Bourgogne, Dijon
  - CHU Grenoble Alpes, La Tronche
  - Hopital Claude Huriez, Lille
  - HCL - Hôpital universitaire de la Croix Rousse, Lyon
  - APHM - Institut Paoli-Calmettes, Marseille
  - CHU de REIMS - Hôpital Robert Debré, Reims
  - Hôpital Hautepierre, Strasbourg
  - CHU de NANCY, Vandœuvre-lès-Nancy

REFERENCES:
- [Result] Doussot B, Doussot A, Ayav A, Santucci N, Deguelte S, Sow AK, El Amrani M, Duvillard L, Piessen G, Girard E, Mabrut JY, Garnier J, Ortega-Deballon P, Fournel I, Facy O. Diagnostic Accuracy of Lipase as Early Predictor of Postoperative Pancreatic Fistula: Results from the LIPADRAIN study. Ann Surg Open. 2024 Sep 11;5(3):e492. doi: 10.1097/AS9.0000000000000492. eCollection 2024 Sep. PMID 39310332